CLINICAL TRIAL: NCT01952873
Title: Rapid Inflation/Deflation Compared With Prolonged High-Pressure Balloon Inflation on the Results of Stent Deployment
Brief Title: Rapid Inflation/Deflation Compared With Prolonged High-Pressure Balloon Inflation
Acronym: INFLATION/DE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 287332
Record Dates: First submitted 2013-09-18; First posted 2013-09-30 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Coronary Stent Occlusion
Keywords: stents; angioplasty, balloon, coronary; coronary artery stenosis; optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid (Active Comparator): The rapid inflation method will consist of reaching an operator determined high-pressure (16 atm) with the stent-deployment balloon and maintaining it the duration of time determined by the operator but <30 sec if the balloon is fully inflated and longer only if the balloon requires a longer duration to become fully inflated.
  Interventions: Other: Rapid inflation
- Prolonged (Experimental): Prolonged inflation will be performed at high pressure(16 atm)and maintained for 30 sec with <0.3 atm drop during that period.
  Interventions: Other: Prolonged inflation

INTERVENTIONS:
Other: Prolonged inflation — Prolonged inflation will be performed at high pressure(16 atm)and maintained for 30 sec with <0.3 atm drop during that period.
  Arms: Prolonged
Other: Rapid inflation — The rapid inflation method will consist of reaching an operator determined high-pressure (16 atm) with the stent-deployment balloon and maintaining it the duration of time determined by the operator but <30 sec if the balloon is fully inflated and longer only if the balloon requires a longer duration to become fully inflated.
  Arms: Rapid

SUMMARY:
It is universally accepted that high-pressure balloon inflation is required to most effectively deploy a coronary balloon-expandable stent. However, there is not consensus nor are there any guidelines regarding the method of balloon inflation, particularly the duration of inflation. Underexpansion and strut malapposition after stent deployment are among the most powerful predictors for adverse vessel outcomes. High-pressure inflation for stent deployment is effective to optimally expand the stent, but unlike in vitro testing in air, there are poorly distensible plaque elements that may not instantaneously yield to the balloon pressure. However, these elements may ultimately yield to prolonged inflation. Most clinical interventional cardiologists inflate for a relatively short period (15-30 sec). The investigators have noted that when balloon pressure is maintained at a certain pressure level it tends to decrease over time, and may require 60-180 or more seconds to maintain pressure stability. This finding implies that plaque elements are yielding slowly over time to the increased pressure, thus increasing expansion, and suggests that a prolonged inflation until balloon pressure stabilizes is more effective than a rapid inflation/deflation sequence to fully expand and appose the stent to the vessel wall. At present there is no consensus on stent deployment strategy. It is our hypothesis that prolonged inflation is superior to the more commonly used strategy of rapid inflation/deflation.

Optimal coherence tomography (OCT), a novel technology that measures near-infrared light reflections and translates them into a 2D image, has an axial resolution nearly 10-times that of intravascular ultrasound (IVUS). Thus it is possible to examine the extent of stent malposition and stent expansion using this modality.

The current randomized trial tests the hypothesis that prolonged balloon inflation until a stable balloon pressure is maintained is more effective than a rapid inflation/deflation sequence when performed to the same balloon inflation pressure.

DETAILED DESCRIPTION:
The rapid inflation method (termed rapid) will consist of reaching a high-pressure (16 atmospheres)with the stent-deployment balloon and maintaining it the duration of time determined by the operator but <30 sec if the balloon is fully deflated and longer only if the balloon requires a longer duration to become fully inflated. Based on previous data, the average time will likely be in the 20-30 sec range. Prolonged inflation (termed prolonged) will be performed at high pressure (16 atmospheres) and maintained for 30 sec with <0.3 atmospheres drop during that period. For example, in the case of 16 atmospheres, the prolonged inflation will require a steady pressure of 15.8-16 atmospheres for at least 30 sec. If the inflation pressure falls 0.3 further pressure will be applied using the digital inflation device until it is again at the target pressure, resetting the 30 second clock. It should be emphasized that if at any time during prolonged inflation there is hemodynamic or electrocardiographic instability, the balloon will be deflated. Based on our previous experience we do not anticipate any safety issues; however, we will measure safety parameters as noted below. After either the rapid or prolonged inflation, an OCT run will be performed to delineate stent expansion and strut apposition. Should the operator determine that the OCT appearance of the stent is unsatisfactory, it is left to the operator to proceed as clinically required, using any further approaches, as he or she sees fit. The results of any further intervention, however, will not be included as part of the data analysis. The study period consists of randomization through the end of the coronary intervention within the catheterization laboratory, for both the efficacy and safety endpoint. The study period will be monitored continuously by a research coordinator and an investigator. All adverse events as described under Safety end points will be reported to the Institutional Review Board (IRB) as per the IRBs prescribed time frame.

ELIGIBILITY:
Inclusion Criteria:

Patients >18 years old with coronary disease with clinical indication for single stent placement in a lesion with a 2.5-3.5 mm diameter and who require OCT for determination of effective stent placement .

Exclusion Criteria:

1. ST segment elevation myocardial infarction 2. Chronic total occlusion 3. Bifurcation lesion or major side branch (>2.5 mm) within the stented area 4. Need for overlapping stents 5. Clinical instability including cardiogenic shock 6. Inability to give informed consent 7. Chronic kidney disease with serum creatinine >1.8 mg/dL 8. Unprotected left main stenosis

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of unopposed stent struts | Day 1 Within first hour after after stent deployment
  How many stents are unopposed
Minimal luminal stent area | Day 1 Within first hour after after stent deployment
  Minimal area of the luminal stent area measured
Minimal lumen stent diameter | Day 1 Within first hour after after stent deployment
  Diameter measured

SECONDARY OUTCOMES:
Number of unopposed stent struts/mm of stent | Day 1 Within first hour after stent deployment
  How many unopposed stent struts are involved
% of patients with complete stent apposition | Day 1 Within first hour after stent deployment
  percentage of patients measured that have a complete stent apposition
Symptomatic ischemia requiring balloon deflation | Intra-procedure
  ischemia requiring balloon deflation
Serious arrhythmia | Intra-procedure and first hour post-Percutaneous Coronary Intervention (PCI)
  Serious arrhythmia during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Barry F Uretsky, M.D., Principal Investigator — Central Arkansas Veterans' Healthcare System
Locations (1):
- John L. McClellan Memorial Veterans Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IPD) sharing plan at this time as the study has been placed on hold.

REFERENCES:
- [Background] Cook JR, Mhatre A, Wang FW, Uretsky BF. Prolonged high-pressure is required for optimal stent deployment as assessed by optical coherence tomography. Catheter Cardiovasc Interv. 2014 Mar 1;83(4):521-7. doi: 10.1002/ccd.24724. Epub 2013 Feb 21. PMID 23436559